CLINICAL TRIAL: NCT02256839
Title: Evaluation of the 4th Generation QuantiFERON-TB Gold Test (CST001) for the Detection of Tuberculosis Infection
Brief Title: Evaluation of the QuantiFERON-TB Test.
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CST001_USA4
Record Dates: First submitted 2014-09-29; First posted 2014-10-06 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- non TB infection: Group tested with CST_001
  Interventions: Device: CST_001
- low exposure risk: Group tested with CST_001
  Interventions: Device: CST_001

INTERVENTIONS:
Device: CST_001

SUMMARY:
To compare the results of the investigational test to the currently approved QuantiFERON-TB Gold In-Tube test.

DETAILED DESCRIPTION:
To compare the specificity of the CST001 assay to the QFT Gold Test in low TB exposure risk subjects and non-tuberculosis mycobacterial infections.

ELIGIBILITY:
Low-exposure Risk Group

Inclusion Criteria:

* No identified risk factors for TB infection

Exclusion Criteria:

* Age less than 18 years or greater than 80 years
* Identified Risk Factors For TB Infection

Non-tuberculous mycobacterial infection Group

Inclusion Criteria:

* history of nontuberculous mycobacterial disease (pulmonary or extrapulmonary) in accordance with the 2007 ATS/IDSA criteria

Exclusion Criteria:

* Age less than 18 years or greater than 80 years
* Identified Risk Factors For TB Infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have either low-exposure rist to tuberculosis or have non-tuberculous mycobacterial infections
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Winthrop, MD, M.P.H, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Sciences University, Portland, Oregon, United States

REFERENCES:
- [Background] QuantiFERON - TB Gold Package Insert (Doc. No. US05990301L). March 2013. Cellestis Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the TB low risk cohort, 2 samples were excluded due to sample transport issues and the third sample for being misdiagnosed as low risk. For the non-TB cohort,1 sample was excluded due to a sample transport issue, and second excluded sample was inadvertently enrolled twice.
Groups:
- Non TB Infection: Non TB Infected Group tested with CST001
- Low Exposure Risk: Low exposure Risk Group tested with CST_001
  CST_001
Period: Overall Study
Arm/Group | Non TB Infection | Low Exposure Risk
Started | 53 | 215
Completed | 51 | 212
Not Completed | 2 | 3
Not completed — Did not meet Eligibility Criteria | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Non TB Infection: Non TB Infected Group tested with CST_001
  CST_001
- Total: Total of all reporting groups
Arm/Group | Non TB Infection | Low Exposure Risk | Total
Number analyzed (Participants) | 51 | 212 | 263
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 207 | 234
  >=65 years | 24 | 5 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 157 | 169
  Male | 39 | 55 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 10 | 11
  Not Hispanic or Latino | 50 | 193 | 243
  Unknown or Not Reported | 0 | 9 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 13 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 49 | 177 | 226
  More than one race | 1 | 13 | 14
  Unknown or Not Reported | 0 | 6 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 212 | 263

OUTCOME MEASURES:

1. Primary Outcome: Clinical Specificity of the CST001 Assay as Measured by the Number of Correctly Identified Actual Negatives
Description: To compare the clinical specificity of the CST001 assay to the QuantiFERON-TB Gold test in low TB exposure risk subjects and non TB infected subjects based on an assessment of known risk factors. These subjects had no identified risk factors of TB infection.
Time Frame: 1 day (At time of enrollment)
Measure: Count of Participants; unit: Participants
Groups:
- Non TB Infection; Low Exposure Risk: Group tested with CST_001
  CST_001
Arm/Group | Non TB Infection | Low Exposure Risk
Number analyzed (Participants) | 51 | 212
Participants | 49 | 208
Statistical Analysis 1: Comparison: Low Exposure Risk; Test type: Equivalence — A 2x2 contingency table with 95% CI; 2 x 2 contingency table = 98.1, 95% CI 2-sided [95.3 to 99.3]
Statistical Analysis 2: Comparison: Non TB Infection; Test type: Equivalence — A 2x2 contingency table with 95% CI; 2 x 2 contingency table = 96.1, 95% CI 2-sided [85.4 to 99.3]

ADVERSE EVENTS:
Groups:
- Low Exposure Risk: Low exposure Risk Group tested with CST001
Arm/Group | Non TB Infection | Low Exposure Risk
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/212
Other Adverse Events (participants affected / at risk) | 0/51 | 0/212

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No